CLINICAL TRIAL: NCT00764114
Title: Comparison of Two Antimicrobial Therapy Duration (6 Weeks Versus 12 Weeks)for Spondylodiscitis
Brief Title: Comparison of Two Antimicrobial Therapy Duration for Spondylodiscitis
Acronym: DTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P050607-AOM05031
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2011-02

CONDITIONS: Vertebral Osteomyelitis
Keywords: Spondylodiscitis; Duration treatment; Antibiotic; men or women more than 18 years; proved bacterial spondylodiscitis; patient for which is decided a treatment antibiotic; the diagnosis on clinical; Radiological; microbiological criteria
MeSH Terms: conditions — Discitis; Multiple Endocrine Neoplasia Type 1 | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): - group A : during 6 weeks after the inclusion
  Interventions: Drug: antibiotic
- 2 (Active Comparator): -group B : during 12 weeks after the inclusion
  Interventions: Drug: antibiotic

INTERVENTIONS:
Drug: antibiotic — 6 or 12 weeks

SUMMARY:
Duration of antimicrobial therapy for spondylodiscitis is not standardized; it could vary from 6 weeks to several months depending on the medical habits. The study hypothesis is that a 6 weeks antimicrobial therapy is not inferior to a 12 weeks.

We run a prospective multi-centric, non inferiority open label trial, randomised in two parallel groups.

The main objective is to compare the efficacy of two durations of antibiotherapy, 6 weeks versus 12 weeks, on the rate of cure in this indication.

The study concerns 400 patients more than 18 years, 70 centres in France are involved.

The duration of the study is 4 years.

DETAILED DESCRIPTION:
In France, incidence of spondylodiscitis is between 1000 and 1500 new cases a year. Micro-organisms mainly in cause are: Staphylococcus aureus, negative coagulase Staphylococcus, Gram negative bacilli and Streptococci; more rarely mycobacteria or Brucella. Actually, optimal duration of antimicrobial therapy is unclear. The rate of cure varies, according to studies, from 90 to 100 % whatever the responsible germ involved. If a 6 weeks antimicrobial therapy duration is not inferior to 12, this would allow to shortening usual antimicrobial therapy duration, and improve tolerance of the treatment, with ecological and economic benefits, following a politics of good use of antibiotics, defined in the French circular n°2002-272 of 02/05/02.

The main objective is to compare two durations of antimicrobial therapy, 6 weeks versus 12 weeks, on the rate of cure of the bacterial spondylodiscitis. Secondary objectives are to compare, according to the duration of treatment antibiotic, 1) Rachidial pain by clinical examination and an analogical visual scale (EVA), 2) Quality of life by the score EQ-5D, 3) Treatment tolerance. 4) Risk factors for failure.

Type of the study is Prospective multi-centric, open label trial, randomised in two parallel groups with direct individual profit.

Antimicrobial therapy is chosen by the physician on charge of the patient according to the germ and to the consensual recommendations.

The study concerns 400 patients.

Inclusion criteria are : men or women more than 18 years, having a proved bacterial spondylodiscitis (not mycobacteria, not fungal nor Brucella), for which an antimicrobial therapy is needed; for the women in age to procreate use of an effective contraception with protected sexual relations and negative pregnancy test (b HCG) is necessary.

Non Inclusion criteria are: infection with no bacteriological identification or mycobacteria, fungal or brucellosis infection, presence of material or recurrence of spondylodiscitis.

Main criterion of evaluation: percentage of success in 1 year defined by the absence of infection : absence of clinical, biological and radiological signs of infection (pain, fever) ; or relapse with the same germ.

This criterion will be estimated beyond the first 6 weeks of treatment antibiotic after the introduction of the treatment and until 1 year after the stop of the treatment. The criteria of the bacteriological diagnosis will be the same.

Design of the study: patients after information consent signed are include and randomised in one arm. They are regularly follow (at 1, 2, 3, 6 and 12 weeks after the beginning of antimicrobial therapy, then at 6 and 12 month after the end of antimicrobial therapy) , with physical examination, biological tests and radiological acts.

The randomisation is centralized, balanced by block, stratifies by centres. (70 centres) The previous duration of the study is of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* men or women more than 18 years
* proved bacterial spondylodiscitis due to pyogenic germ (no mycobacteria, no fungus or brucella), for which is decided a treatment antibiotic
* diagnosis is based on clinical,radiological and microbiological criteria
* women in age to procreate, use of an effective contraception with protected sexual relations and negative pregnancy test (b HCG).

Exclusion Criteria:

* infection with no bacteriological identification
* infection due to mycobacteria, brucella or fungus
* presence of material
* recurrence of spondylodiscitis
* Patient whose life expectation is 1-year-old subordinate
* pregnant or breast-feeding Woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2006-11; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percentage of success in 1 year defined by the absence of infection : absence of clinical, biological and radiological signs of infection (pain, fever) ; or relapse with the same germ. | 1 year after the stop of the treatment.

SECONDARY OUTCOMES:
1)Effective antibiotherapy duration | 12 months
2) Failure rate at 6 month | 6 months
3)Rachidial pains (clinical examination and analogical visual scale of the pain) at every visit | 6 an 12 month
4)Quality of life by the score EQ-5D at 6 and 12 month | 6 and 12 month
5)Observance of the treatment measured at every visit | 6 and 12 month
6)Appearance of microbial resistances estimated by comparison of antibiogram in case of failure | during 12 months
7)Antimicrobial therapy tolerance measure at each visit | 6 and 12 month
8)Identification of risk factors for failure | during 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bernard, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Chu Raymond Poincare, Garches, France

REFERENCES:
- [Derived] Desoutter S, Cottier JP, Ghout I, Issartel B, Dinh A, Martin A, Carlier R, Bernard L; Duration of Treatment for Spondylodiscitis Study Group. Susceptibility Pattern of Microorganisms Isolated by Percutaneous Needle Biopsy in Nonbacteremic Pyogenic Vertebral Osteomyelitis. Antimicrob Agents Chemother. 2015 Dec;59(12):7700-6. doi: 10.1128/AAC.01516-15. Epub 2015 Oct 5. PMID 26438497
- [Derived] Zervou FN, Zacharioudakis IM, Mylonakis E. ACP Journal Club. 6 weeks of antibiotics was noninferior to 12 weeks for clinical cure in pyogenic vertebral osteomyelitis. Ann Intern Med. 2015 May 19;162(10):JC7. doi: 10.7326/ACPJC-2015-162-10-007. No abstract available. PMID 25984880
- [Derived] Bernard L, Dinh A, Ghout I, Simo D, Zeller V, Issartel B, Le Moing V, Belmatoug N, Lesprit P, Bru JP, Therby A, Bouhour D, Denes E, Debard A, Chirouze C, Fevre K, Dupon M, Aegerter P, Mulleman D; Duration of Treatment for Spondylodiscitis (DTS) study group. Antibiotic treatment for 6 weeks versus 12 weeks in patients with pyogenic vertebral osteomyelitis: an open-label, non-inferiority, randomised, controlled trial. Lancet. 2015 Mar 7;385(9971):875-82. doi: 10.1016/S0140-6736(14)61233-2. Epub 2014 Nov 5. PMID 25468170